CLINICAL TRIAL: NCT06991699
Title: A Novel Digitally Driven Approach for Gummy Smile Solution Using Milled Sub-nasal Stent: A Clinical Study
Brief Title: A Novel Digitally Driven Approach for Gummy Smile Solution Using Milled Sub-nasal Stent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: taher helmy ismail metwaly (Other)
Responsible Party: Sponsor-Investigator, taher helmy ismail metwaly, MSc. Candidate of Periodontology, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3/1-2024
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Gummy Smile

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Milled PEEK Stent (Experimental)
  Interventions: Other: Milled PEEK Stent

INTERVENTIONS:
Other: Milled PEEK Stent — A CBCT will be performed to assess the anatomy of the subnasal area and plan the position, size, shape and thickness of the PEEK Stent. These data will be transferred to a 3D planning software to generate a digital model. Eventually, the PEEK stents will be milled in a milling machine and sterilized in ethylene oxide before the surgery. Local anesthesia will be administered into the vestibular mucosa along the extension of the anterior maxilla. VISTA technique begins with a vestibular access incision in the midline frenum and 2 bilateral incisions at premolar area. A periosteal elevator will be introduced through the incision and inserted between the bone and periosteum to elevate the tissue, creating a subperiosteal tunnel, extending distally based on the dynamic of the smile. The PEEK stent will be in one piece. They will be placed onto the bone and stabilized with 2 bone graft screw for each side. The midline incision and the lateral incisions will be sutured primarily.

SUMMARY:
The objective of this study is to assess the effectiveness of a Polyether ether ketone (PEEK) stent for management of gummy smile.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals
* Chiefs complain gummy smile
* Gummy smile due to short hypermobile upper lip
* Gingival Display not more than 5 mm

Exclusion Criteria:

* Pregnancy
* Lactation
* History of smoking more than 10 cigarettes per day
* Systemic conditions or intake of medications that could affect soft and hard tissue healing
* Use of orthodontic appliances
* Gingival display above 5mm

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Gingival display | up to 6 months
  Distance from gingival margin to lower border of upper lip vermilion border will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt